CLINICAL TRIAL: NCT02063048
Title: The Comparative Effectiveness of Clinic-Based Weight Loss Strategies
Brief Title: Text Messaging for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Center for Health Systems Research at Denver Health (Unknown); Colorado Health Outcomes Program (Other)
Responsible Party: Principal Investigator, Henry Fischer, Physician - Internal Medicine, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-1606 (Fischer); 1R24HS022143-01 (AHRQ)
Record Dates: First submitted 2014-02-10; First posted 2014-02-14 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Body Weight; Body Weight Changes; Prediabetic State; Prediabetes
Keywords: weight loss; Text Messaging; Short Message Service; Text Messages
MeSH Terms: conditions — Body Weight; Body Weight Changes; Prediabetic State; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care for Weight Loss (No Intervention): Patients randomized to this arm will not receive text messages or any other weight-loss support besides usual care provided at Denver Health. They will receive a weight loss educational packet and be asked to follow up with their primary care provider to further discuss their efforts at weight loss with additional follow-up as directed by their provider. They will be contacted periodically to be weighed. Providers will not be made aware that their patients are participating in the study's control arm.
- Text Message Based Weight Loss Support (Experimental): Patients will receive the same weight loss educational packet as those randomized to usual care. Patients will be assisted in choosing a self-management goal related to exercise and to eating behaviors. They will receive text messages at a frequency up to 1x daily; input from focus groups will guide text message frequency.
  Interventions: Behavioral: Text Message Based Weight Loss Support

INTERVENTIONS:
Behavioral: Text Message Based Weight Loss Support
  Arms: Text Message Based Weight Loss Support

SUMMARY:
The purpose of this study is to compare the effectiveness of text message-based support to usual care at promoting weight loss in patients with pre-diabetes.

DETAILED DESCRIPTION:
Text messaging has been shown to be effective for weight-loss in very limited testing. DH has experience with both text message based intervention and weight management intervention. This study aims to enhance Denver Health's (DH) existing Patient Relationship Management (PRM) text message (SMS) infrastructure to include culturally-appropriate outreach to promote weight loss.

Subjects will be randomized into one of two arms:

* Usual care: Patients randomized to this arm will not receive text messages or any other weight-loss support besides usual care provided at DH. They will receive a weight loss educational packet and be asked to follow up with their primary care provider to further discuss their efforts at weight loss with additional follow-up as directed by their provider. They will be contacted periodically to be weighed. Providers will not be made aware that their patients are participating in the study's control arm.
* Text Message-based weight loss support. Patients will receive the same weight loss educational packet as those randomized to usual care. Patients will be assisted in choosing a self-management goal related to exercise and to eating behaviors. They will receive text messages at a frequency up to 1x daily; input from focus groups will guide text message frequency.

SMS content is similar to the Diabetes Prevention Program (DPP) curriculum and will fall into the following categories:

* Outgoing "tips of the day"
* Interactive messages that solicit a simple response for the day from the participant
* Outgoing reminders to inform participant about events in the community and about clinic appointments with their primary care provider.

Basic descriptive statistics for categorical variables will be generated to describe the baseline demographic and clinical characteristics. Univariate analyses will be performed to determine whether there are differences between patients in the three arms of the intervention. For clinical outcomes, general linear mixed effects models will be used with intervention and time (and their interactions) specified as fixed effects to determine whether change over time in outcomes differs significantly for the three groups. A random subject effect will be specified to model the correlation of observations taken on an individual. Contrasts will be constructed to test the difference in interventions at six months and 12 months. If the data do not follow an approximate normal distribution or cannot be normalized using log transformation the ranks of the outcomes will be analyzed in the mixed effects model. All statistical analyses will be performed using Statistical Analysis Software (SAS) version 9.2.

The study is powered to detect a difference at six months between the text message group and the usual care group. Previous research suggests that, with 60 participants per group, researchers would have 89% power to detect a difference between groups of 1.7 kg. The investigators think that this is a reasonable estimate, as subjects in the control group in this study lost 0.4 kg, and it is believed that subjects in the control group will be weight stable. While investigators anticipate that patients who participate in the DPP program will lose weight, it is believed participation across the usual care and SMS groups will be comparable as i) randomization is stratified to the two groups by past participation in the DPP and ii) relatively equal participation in the two groups is anticipated throughout the intervention period. This stratification is intended to equalize the effects of class-attendance heterogeneity across the two study groups. The study aims to have 90 participants per group to improve the power for sub-group analyses.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age or older
* Ownership of a cell phone with SMS capabilities
* HbA1c greater than 5.6 but less than 6.5
* BMI ≥ 25 kg/m2 and less than 50 kg/m2
* English or Spanish speakers.

Exclusion Criteria:

* Individuals with co-morbid illness with life expectancy less than 12 months (e.g., terminal cancer, Child's Class C hepatic cirrhosis)
* Diabetes based on an ICD-9 code in previous 3 years
* Institutionalized individuals
* Individuals not planning to stay in the area at least 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Absolute weight loss in pounds | 12 months
  Outcomes will be analyzed at baseline and at 6-month and 12-month follow-ups.

SECONDARY OUTCOMES:
Percent weight loss | 12 months
  Outcomes will be analyzed at baseline and at 6-month and 12-month follow-ups.
Change in glycemic control as measured by HbA1c and fasting glucose | 12 months
Patient Engagement Measures | 12 months
  Response rate to text message prompts
Percent of patients who maintain or lose weight | 12 months
  defined as weight gain less than two pounds
Changes in systolic and diastolic blood pressure | 12 months
  based on usual care measurements
Change in LDL-cholesterol | 12 months
  based on usual care measurements
Operating costs per participant receiving intervention | 12 months
  Costs from the perspective of the health system, including all personnel costs and technology costs, will be calculated. The upper 2.5% of the cost distribution curve will be truncated to eliminate outliers that would artificially skew results and use non-parametric methods if the distribution is non-normal as expected. The effect of scaling the intervention up two-fold and five-fold will undergo sensitivity analyses.
Patient Engagement Measures | 12 months
  Acceptability of the text-message based approach through individual interviews

CONTACTS AND LOCATIONS:
Overall Officials: Henry Fischer, MD, Principal Investigator — Denver Health; Edward Havranek, MD, Study Director — Denver Health
Locations (1):
- Denver Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Fischer HH, Pereira RI, Moore SL, Durfee MJ, Rozwadowski JM, Havranek EP. Response to Comment on Fischer et al. Text Message Support for Weight Loss in Patients With Prediabetes: A Randomized Clinical Trial. Diabetes Care 2016;39:1364-1370. Diabetes Care. 2016 Nov;39(11):e207-e208. doi: 10.2337/dci16-0024. No abstract available. PMID 27926904
- [Derived] Fischer HH, Fischer IP, Pereira RI, Furniss AL, Rozwadowski JM, Moore SL, Durfee MJ, Raghunath SG, Tsai AG, Havranek EP. Text Message Support for Weight Loss in Patients With Prediabetes: A Randomized Clinical Trial. Diabetes Care. 2016 Aug;39(8):1364-70. doi: 10.2337/dc15-2137. Epub 2016 Feb 9. PMID 26861922